CLINICAL TRIAL: NCT07248800
Title: Effect of Tele-dentistry on Awareness of Egyptian Children and Caregivers Regarding Risks of Early Childhood Caries; Prospective Cohort Study
Brief Title: Oral Health Awareness Among Egyptian Population
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelhameed Hamid Mohammad Hijazi, Lecturer, Sinai University
Other Study IDs: SU.REC.2024 (24 H)
Record Dates: First submitted 2025-11-16; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Early Childhood Caries (ECC); Oral Health Behavior Change

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kindergarten children

SUMMARY:
The objective of this research is to investigate the effect of digital tele-dentistry application using AI-generated content on the awareness and performance among a sample of Egyptian children and their caregivers in both kindergarten and pediatrician offices.

● Aim of the study The aim of the current study is to evaluate the use of teledentistry in the field of public health enhancement and monitoring, especially for children's oral health.

ELIGIBILITY:
Inclusion Criteria:

* Parents and caregivers of children aged 5 - 10 years old of any gender

Exclusion Criteria:

* 1- Children <5 years old or >10 years old 2- Children with special needs, including:

  1. Physical disability (sensory or motor defects)
  2. Mental retardation 3- Uncooperative children or caregivers

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and caregivers in Ismailia governorate are visiting kindergartens and pediatric clinics.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Awareness level | 6 months
  awareness and performance change after using tele-dentistry to enhance oral health measures and screening, using an evaluation form about dietary habits and dental hygiene practices were registered by the children and their caregivers daily during the trial period
  1. The baseline awareness level was recorded (pretest), using four domains-based questionnaires about oral health and healthy diet practices, risk factors for early childhood caries and enamel demineralization will be given to the caregivers and parents of recruited children.
  2. Awareness level was assessed after the end of one month exposure using the same questionnaire, repeated after 3 month and post-trial after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No